CLINICAL TRIAL: NCT00013273
Title: Physical Conditioning in Management of Chronic Venous Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1792R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Venous Insufficiency
Keywords: Venous insufficiency, plethysmography, hypertension
MeSH Terms: conditions — Venous Insufficiency; Hypertension | interventions — Exercise Therapy

INTERVENTIONS:
Procedure: Physical Conditioning

SUMMARY:
The purpose of this research is to evaluate the efficacy of a structured program of physical therapy in ameliorating the adverse consequences of Chronic Venous Insufficiency (CVI). The study will also investigate the interrelationship among measure of chronic venous diseases: lower limb muscle strength, mobility, and other symptoms of CVI important to the quality of life. Sixty patients will be randomized to a 6 months physical therapy program or to a control group.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate the efficacy of a structured program of physical therapy in ameliorating the adverse consequences of Chronic Venous Insufficiency (CVI). A secondary purpose is to investigate the interrelationship among measure of chronic venous diseases: lower limb muscle strength, mobility, and other symptoms of CVI important to the quality of life. Sixty patients will be randomized to a 6 months physical therapy program or to a control group. All subjects will undergo a complete hemodynamic and psychiatric assessment. Key measures will be repeated twice to quantify trend and stability of the baseline measures. Skin biopsies will be obtained in selected patients who demonstrate a response to the physical therapy to evaluate the ultrastructural response therapy. Physical therapy will be conducted 1-3 times per week. Participants will be visited at home and a program will be tailored for each individual to maximize compliance. Validated, standardized questionnaires (FIM, SF-36, OARS, CHART) and functional ratings will be employed at commencement,3,6 and 12 months. Evaluations of hydrodynamics, muscle strength, and ankle motion will be conducted monthly during active physical therapy. Participants in active therapy will be offered to wait listed control group after 6 months.

ELIGIBILITY:
Patients with severe form of chronic venous insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1999-01; Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D. Assistant Director — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Wijegupta Ellepola, Program Analyst — Program Analysis and Review Section (PARS), Rehabilitation Research and Development Service
Locations (1):
- VAMC, East Orange, NJ, East Orange, New Jersey, United States